CLINICAL TRIAL: NCT07033858
Title: Investigating the Effect of Low-dose Extended-release Tacrolimus and Sirolimus on the Short-term Outcomes of Allograft Kidney Transplantation
Brief Title: Evaluaion the Short Term Effects of Advograf Plus Rapamiune After Kidney Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, assistant professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBMU-1404-2
Record Dates: First submitted 2025-05-27; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Kidney Transplant; Complications
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Advograf plus Cellcept plus Prednisolone
- Intervention (Other): Advograf plus Rapamiune plus Prednisolone
  Interventions: Drug: Rapamune Pill

INTERVENTIONS:
Drug: Rapamune Pill — Rapamiune Tablet 1mg daily plus Advograf plus prednisolone
  Other Names: Sirolimus
  Arms: Intervention

SUMMARY:
Cornerstone immunosuppressive therapy currently relies on immediate-release tacrolimus, a calcineurin inhibitor (CNI) that is potentially nephrotoxic and is more diabetogenic than cyclosporine A. A new formulation of tacrolimus has been launched: an extended-release formulation (Advagraf®/Astagraf XL®, Astellas company).

DETAILED DESCRIPTION:
This study wants to assess the efficacy of an extended-release formulation of tacrolimus (Advagraf®/Astagraf XL®) used in conjunction with an mTOR-inhibitor agent (sirolimus ) instead of MMF to evaluate the hypothesis that this regimen is associated with good allograft outcome, and might also prevent late-onset cytomegalovirus infection. Advagraf®-based immunosuppression given to de novo kidney-transplant recipients may also increase patients' adherence to treatment due to once-daily usage of the drug.

ELIGIBILITY:
Inclusion Criteria:

* All Kidney transplant recipients

Exclusion Criteria:

* Kidney-Pancreas transplant BMI>30 cPRA>0%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Kidney function | through study completion, an average of 1 year
  gfr measurement
Post-transplant viral Infections | through study completion, an average of 1 year
  Number of participents with positive blood tests of CMV and BK as assessed by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Dalili, Principal Investigator — SBMU
Locations (1):
- Nooshin Dalili, Tehran, Iran